CLINICAL TRIAL: NCT02699346
Title: An Open-Label, Non-Randomized Study Designed to Evaluate the Correlation of HS-1000 Device Capabilities in the Diagnosis and Assessment of Patients After Concussion With Clinical Evaluation
Brief Title: An Evaluation of HS-1000 Device Capabilities in the Diagnosis and Assessment of Patients After Concussion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HeadSense Medical (Industry)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-010
Record Dates: First submitted 2016-02-26; First posted 2016-03-04 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Brain Concussion; Brain Injuries
Keywords: concussion; mild traumatic brain injuries
MeSH Terms: conditions — Brain Concussion; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HS-1000 recording (Experimental): Eligible patients and healthy subjects will be enrolled into the study and HS-1000 headset portion of the device will be placed in their ears. HS-1000 monitoring intervals will last from 20 minutes continuously. Following completion of data collection, HS-1000 will be removed.
  Interventions: Device: HS-1000 recording

INTERVENTIONS:
Device: HS-1000 recording

SUMMARY:
The HeadSense (HS) HS-1000 device, a new non-invasive brain monitor is expected to safely and accurately monitor concussed patients with minimal discomfort, potentially providing a new modality for concussion measurement. The device is based on advanced signal analysis algorithms that analyze a very low frequency acoustic signal (within the audible range) generated by the device. The acoustic signal is transmitted using a small transmitter, placed in the participant's ear, and picked by an acoustic sensor placed in the other ear.

DETAILED DESCRIPTION:
Concussion diagnosis and assessment suffers from lack of a gold-standard measurement, leaving physicians to rely on physical and neurological examinations, neurocognitive/mental status testing, and balance examination, which can be time-consuming and influenced by subjective factors. In order to address this significant drawback, there is a need for novel modalities that diagnose and monitor concussion in a quick easy-to-use and non-invasive manner.

Based on our previous analysis of the physiological processes using acoustic signals that were collected and analyzed so far, our hypothesis is that the HS-1000 is capable of diagnosing and monitoring concussed patients, based on the acoustic raw data derived from the generated acoustic signal along with the analysis of the acoustic signals that derive from the physiological processes in the brain. These processes, e.g. cerebral blood-flow and the respiratory cycle, are impaired during changes in intracranial pressure (ICP) and are hypothesized to change as well once the patient is concussed.

Concussed athletes will be identified through routine visits at the Vanderbilt Sports Concussion Center. Controls will be identified among non-concussed athletes being seen at Vanderbilt Sports Medicine and will be offered participation.

After signing informed consent, both healthy subjects and patients will undergo screening assessments for this study. Eligible patients and healthy subjects will be enrolled into the study and HS-1000 headset portion of the device will be placed in their ears. HS-1000 monitoring intervals will last from 20 minutes continuously. Following completion of data collection, HS-1000 will be removed.

Safety evaluation will include monitoring of adverse events throughout the study.

The study duration for each patient will be up to 1 hour. Healthy subjects will undergo two recordings approximately two weeks apart.

Post-concussion patients will have multiple sessions:

* Session #1 Baseline recording as soon as possible
* Session #2 48 hours after session #1
* Session #3 1 week after session #1
* Session #4 1 month after session #1

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with no previous concussions:

  1. Male or female subjects, aged 13 - 25 years old at screening visit
  2. Subjects who were previously diagnosed by standard methods as healthy subjects with no previous concussions
  3. Subject is able and willing to comply with the requirements of the protocol
  4. Subject is able to understand and sign written informed consent to participate in the study
* Post-concussion diagnosed patients:

  1. Male or female subjects, aged 13-25 years at screening visit
  2. Subjects who were previously diagnosed by standard methods as suffering from concussion
  3. Subject is able and willing to comply with the requirements of the protocol
  4. Subject is able to understand and sign written informed consent to participate in the study

Exclusion Criteria:

1. Local ear infection
2. Known allergy or hypersensitivity to any of the test materials or contraindication to test materials
3. Subjects currently enrolled in or less than 30 days post-participation in other investigational device or drug study(s), or receiving other investigational agent(s)
4. Any condition that may jeopardize study participation (e.g., abnormal clinical or laboratory finding) or interpretation of study results, or may impede the ability to obtain informed consent
5. History of psychiatric illness, chemical dependency, Attention-Deficit Hyperactivity Disorder (ADHD), Learning Disability, seizure disorder, prior neurosurgical intervention
6. Current use of psychotropic medication

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-06 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
To measure ICP values by using the HS-1000 in healthy subjects and concussed subjects | 20 minute recording session
Determine the correlation between ICP measurements obtained from the HS-1000 device and the clinical findings from the modified Balance Error Score System (mBESS) and ImPACT scores in post-concussion patients. | 20 minute recording session

SECONDARY OUTCOMES:
To evaluate the ergonomic and functional aspects of using the HS-1000 by having the operators of the device complete a brief 5 question survey about the ease or difficulty in using the device. | 20 minute recording sessin

CONTACTS AND LOCATIONS:
Overall Officials: Allen K Sills, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No